CLINICAL TRIAL: NCT01708694
Title: Role of Slowly Digesible Starch on Diabetes Risk Factors In Pre-diabetic People
Brief Title: Role of Slowly Digesible Starch on Diabetes Risk Factors
Acronym: STARCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Eric Ravussin, Principal Investigator, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: PBRC 12009; R01DK092575 (NIH)
Record Dates: First submitted 2012-10-10; First posted 2012-10-17 (Estimated); Last update posted 2017-12-15 (Actual); Status verified 2017-12

CONDITIONS: Prediabetes
MeSH Terms: conditions — Prediabetic State | interventions — Amylose; Amylopectin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo Starch (Placebo Comparator): Yogurt with about 45 g/day of placebo starch (amylopectin).
  Interventions: Dietary Supplement: Amylose
- Experimental Starch (Experimental): Yogurt with about 45 g/day of slowly digestible starch (amylose).
  Interventions: Dietary Supplement: Amylopectin

INTERVENTIONS:
Dietary Supplement: Amylose — One group of participants will consume a yogurt containing 45 g of amylose (the slowly digesting starch) for 3 months.
  Arms: Placebo Starch
Dietary Supplement: Amylopectin — The second group will consume a yogurt containing 45 g of a different starch called amylopectin (the "placebo") for 3 months.
  Arms: Experimental Starch

SUMMARY:
The purpose of this study is to determine the effect of a slowly digesting starch on gut bacteria, sugar and fat metabolism, hunger hormones, and body fat in people with pre-diabetes.

DETAILED DESCRIPTION:
In a double blind randomized controlled clinical trial, the investigators will test the effect of slowly digesting starch (amylose) versus a placebo starch (amylopectin) on risk factors for type 2 diabetes. For the study, about 95 obese participants (ages 35-65) with pre-diabetes (impaired fasting glucose) will consume a yogurt containing about 45 g of either the experimental or placebo starch daily for 3 months. The investigators will test the hypothesis that, compared to controls, a daily intake of 45 g of amylose for 3 months will improve risk factors for the development of type 2 diabetes (insulin sensitivity and secretion) by decreasing ectopic fat depots and decreasing inflammation in parallel with a change in colonic microbial populations.

ELIGIBILITY:
Inclusion Criteria

* Have a body mass index between 30 and 44.9 kg/m2
* Are 35-65 years of age
* Have pre-diabetes, which means impaired fasting glucose (IFG)
* Are willing to complete nutritional and activity questionnaires and 2-3 weeks of baseline testing
* Are willing to enroll in the 3-month intervention and maintain the same level of exercise during the study
* Are willing to maintain weight throughout the study

Exclusion Criteria

* Have evidence of cardiovascular disease, diabetes, symptomatic cholelithiasis (gallstones), or cancer
* Have a fasting blood glucose less than 100 mg/dL or greater than 125 mg/dL
* Have an average screening blood pressure > 150/100 mm Hg
* Are a pre-menopausal woman but do not have a regular menstrual cycle
* Are pregnant or breastfeeding
* Chronically use medications including diuretics, steroids, and adrenergic-stimulating agents
* Have emotional problems such as clinical depression or other diagnosed psychological conditions
* Use hormonal contraceptives, oral or parenteral glucocorticoids, or any other medication known to influence glucose or insulin homeostasis (balance), within 1 month of study
* Have a clinically significant gastrointestinal malabsorption syndrome, chronic diarrhea, or use antibiotics within one month of study
* Have abnormal laboratory markers (e.g., elevated potassium levels, hemoglobin or hematocrit below the lower limit of normal)
* Chronically consume alcohol (> 4 servings per day) or actively smoke cigarettes (> 1/4 pack per day)
* Are on any chronic medication that has not had a stable dose for 1 month or longer
* Are required to perform of any kind of heavy physical activity
* Have metal objects in the body, such as a pacemaker, metal pins, bullet, etc.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2012-08; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Insulin Sensitivity and Secretion | 3 months
  Insulin sensitivity and secretion will be assessed via a Frequently Sampled Intravenous Glucose Tolerance Test (FSIGTT).

SECONDARY OUTCOMES:
Body Composition | 3 months
  DXA and MRS will be performed to measure body composition (adipose, muscle, bone mineral content) and to measure hepatic and intramyocellular lipids, respectively.
Gut Microbiota | 3 months
  Stool samples will be collected and fecal bacteria diversity will be measured in conjunction with metagenomic analysis.
Satiety | 3 months
  Satiety hormones will be measured following ingestion of a standardized smoothie (Standard Meal Test). Satiety will be measured through visual analogue scales (VAS), remote food photography, and a food intake test.
Hunger | 3 months
  Hunger will be measured through visual analogue scales (VAS), remote food photography, and a food intake test.

CONTACTS AND LOCATIONS:
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- [Derived] White U, Peterson CM, Beyl RA, Martin CK, Ravussin E. Resistant Starch Has No Effect on Appetite and Food Intake in Individuals with Prediabetes. J Acad Nutr Diet. 2020 Jun;120(6):1034-1041. doi: 10.1016/j.jand.2020.01.017. Epub 2020 Apr 9. PMID 32280055
- [Derived] Peterson CM, Beyl RA, Marlatt KL, Martin CK, Aryana KJ, Marco ML, Martin RJ, Keenan MJ, Ravussin E. Effect of 12 wk of resistant starch supplementation on cardiometabolic risk factors in adults with prediabetes: a randomized controlled trial. Am J Clin Nutr. 2018 Sep 1;108(3):492-501. doi: 10.1093/ajcn/nqy121. PMID 30010698
- [Derived] Marlatt KL, White UA, Beyl RA, Peterson CM, Martin CK, Marco ML, Keenan MJ, Martin RJ, Aryana KJ, Ravussin E. Role of resistant starch on diabetes risk factors in people with prediabetes: Design, conduct, and baseline results of the STARCH trial. Contemp Clin Trials. 2018 Feb;65:99-108. doi: 10.1016/j.cct.2017.12.005. Epub 2017 Dec 21. PMID 29274892